CLINICAL TRIAL: NCT00859079
Title: Efficacy of a Continuous GLP-1 Infusion in Comparison to a Structured Insulin Infusion Protocol to Reach Normoglycemia in Non-Fasted Type 2 Diabetic Patients
Brief Title: Efficacy of GLP-1 Infusion in Comparison to an Insulin Infusion Protocol to Reach Normoglycemia Type 2 Diabetic Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Dr. Thomas Wascher, Medical University of Graz
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: TCW-GLP1-1
Record Dates: First submitted 2009-03-07; First posted 2009-03-10 (Estimated); Last update posted 2009-03-10 (Estimated); Status verified 2009-03

CONDITIONS: Diabetes Mellitus Type 2; Hyperglycemia
Keywords: diabetes mellitus type 2, GLP-1, insulin infusion
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hyperglycemia | interventions — Glucagon-Like Peptide 1; insulin, neutral

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GLP-1 (Active Comparator): Intravenously administered GLP-1
  Interventions: Drug: GLP-1
- Insulin intravenously (Active Comparator): Insulin intravenously according to the Munich registry
  Interventions: Drug: Human regular insulin intravenously

INTERVENTIONS:
Drug: GLP-1 — Patients received GLP-1 intravenously at a dose of 1.2 pmol/kg/min for at maximum 8 hours.
  Other Names: GLP-1 infusion (CLINALFA, Laeufelingen, Switzerland)
  Arms: GLP-1
Drug: Human regular insulin intravenously — Human regular insulin intravenously according to the Munich-registry.
  Other Names: Insulin Actrapid, NovoNordisk, Denmark
  Arms: Insulin intravenously

SUMMARY:
The aim of the investigators study was to compare for the first time efficacy and safety of intravenously administered GLP-1 with an established intravenous insulin regimen in hyperglycaemic type 2 diabetic patients.

DETAILED DESCRIPTION:
Intervention studies in patients with acute myocardial infraction or cardiac surgery, using intravenously administered human insulin, suggest that normalization of hyperglycemia can reduce morbidity as well as mortality in these patients. Insulin-based regimens require frequent blood glucose measurements and adjustments of infusion rate to achieve normoglycemia.

In addition, hypoglycaemia is a frequent and important side effect. Glucagon-Like-Peptide 1 (GLP-1) is an insulinotropic, glucagonostatic gastrointestinal hormone that lowers glucose in a glycemia-dependent manner and therefore does not cause hypoglycemia.

The aim of our study was to compare for the first time efficacy and safety of intravenously administered GLP-1 with an established intravenous insulin regimen in hyperglycaemic type 2 diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus
* Fasting glycemia above 150 mg/dl
* Signed informed consent

Exclusion Criteria:

* Patients with heart failure > NYHA II
* Uncontrolled hypertension
* Impaired kidney function (creatinine > 3 mg/dl)
* Acute infection

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2006-06; Primary Completion 2006-12 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
time to reach a plasma glucose below 115 mg/dl | 0,30,60,120,150,180,210,240,270,300,330,360,390,420,450,480,510 min

SECONDARY OUTCOMES:
plasma glucose after 2 and 4 hours as well as maximum glycemia | 0,30,60,120,150,180,210,240,270,300,330,360,390,420,450,480,510 min
number of hypoglycaemic episodes | 0,30,60,120,150,180,210,240,270,300,330,360,390,420,450,480,510 min

CONTACTS AND LOCATIONS:
Overall Officials: Thomas C Wascher, MD, Principal Investigator — Medical University of Graz, Dept. of Internal Medicine, Auenbruggerpl. 15, 8036 Graz, Austria
Locations (1):
- Medical University of Graz, Department for Internal Medicine, Graz, Austria